CLINICAL TRIAL: NCT06956157
Title: Altered Brain Glutamate Level and Inhibitory Control in Treatment-Resistant Obsessive-Compulsive Disorder After N-acetylcysteine (NAC) Augmentation Therapy
Brief Title: NAC for Treatment-Resistant OCD and Other Related Disorders
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, sunnyrong, Director, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: KY2020-572; 2021A1515011431 (Other Grant/Funding Number: Natural Science Foundation of Guangdong Province)
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Obsessive Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- N-acetylcysteine group (Experimental): NAC (N-Acetylcysteine Tablets, brand name: Flumucil) has a drug specification of 600 mg per tablet. In the first week, participants took 1200mg/d (one tablet three times daily: morning, noon, and evening). Starting from the second week until the end of the 12-week study, they took 3600mg/d (three tablets twice daily: morning and evening).
  Interventions: Drug: N-Acetylcysteine Tablets
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet
- Healthy Control Group (No Intervention)

INTERVENTIONS:
Drug: N-Acetylcysteine Tablets — In addition to participants' existing medication regimens, NAC will be added.
  Arms: N-acetylcysteine group
Drug: Placebo Oral Tablet — Placebo oral tablets are identical in appearance (size, shape, color), packaging, taste, and administration schedule to the N-Acetylcysteine tablets to maintain blinding. The tablets contain inert excipients and no active pharmacological ingredients.
  Arms: Placebo group

SUMMARY:
This is a randomized, double-blind, placebo-controlled study investigating N-acetylcysteine (NAC) as an augmentation therapy for individuals with treatment-resistant obsessive-compulsive disorder (TR-OCD), studied within a broader cohort of treatment-resistant Obsessive-Compulsive and Related Disorders (OCRDs).

The study's primary aim is to investigate the neurobiological mechanism by which NAC improves inhibitory control deficits in TR-OCD. This is achieved by using Magnetic Resonance Spectroscopy (MRS) to measure changes in thalamic glutamatergic metabolism. A secondary aim is to assess the clinical efficacy of this augmentation strategy on symptom severity. The central hypothesis is that improvements in inhibitory control are mediated by NAC-induced changes in brain glutamate levels.

DETAILED DESCRIPTION:
Please note: This study was initially designed to investigate the effects of N-acetylcysteine (NAC) across the broader spectrum of treatment-resistant Obsessive-Compulsive and Related Disorders (OCRDs), including cohorts such as Excoriation (Skin-Picking) Disorder. The overarching scientific objective was to use NAC to elucidate the neurobiological mechanisms underlying inhibitory control deficits in this difficult-to-treat population, and thereby inform the development of novel therapeutic strategies.

Upon completion of recruitment for the current analysis phase and prior to any unblinking, we finalized our analytical strategy. To ensure the primary analysis was adequately powered to yield a definitive conclusion, it was focused on the treatment-resistant OCD (TR-OCD) cohort, which comprised the substantial majority of the sample accrued to date.

Consequently, the TR-OCD cohort was designated as the primary population for the main efficacy and mechanistic analyses. Other OCRD subgroups enrolled under the same protocol were designated for planned secondary and exploratory analyses, in line with their respective sample sizes. Analyses of these subgroups, including the SPD cohort, will be conducted once sufficient data have been accrued for robust statistical testing.

This registration has been updated to accurately and transparently reflect this final, pre-specified analytical plan, ensuring the public record aligns with the study's primary, hypothesis-driven conclusions.

ELIGIBILITY:
1.Inclusion Criteria for Patient:

(1) Age between 12 and 55 years. (2) A primary diagnosis of OCD according to DSM-5 criteria. (3) Excoriation (Skin-Picking) Disorder (SPD) according to DSM-5 criteria.

(4) Met criteria for treatment resistance, defined as: (a) A Y-BOCS score ≥ 16. (b) A history of inadequate response (<25% reduction in Y-BOCS score) to at least two different serotonin reuptake inhibitors (SSRIs) at an adequate dose for at least 12 weeks each.

1.2 Inclusion Criteria for Healthy Controls:

(1) Age and sex-matched to the patient group. (2) No personal history of any psychiatric disorder.

1.3 Exclusion Criteria for All Participants: (1) Presence of any contraindications to 3T MRI scanning (e.g., metallic implants, claustrophobia). (2) Current (within the past 6 months) diagnosis of a substance use disorder. (3) Significant or unstable neurological illness (e.g., epilepsy, multiple sclerosis, brain tumor). (4) History of significant head trauma or neurosurgery.

1.4 Additional Exclusion Criteria for Patients with TR-OCD:

(1) Current or lifetime diagnosis of a primary psychotic disorder (e.g., schizophrenia), bipolar I/II disorder, or intellectual disability. (2) Any contraindication to the use of N-acetylcysteine.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Neurometabolite Concentrations in Key Brain Regions | Baseline, Post-treatment (Week 12)
  Change from baseline to Week 12 in the concentrations of Glutamate (Glu), Glutamate+Glutamine (Glx), and Glutathione (GSH) within two pre-specified regions of interest: the thalamus and the anterior cingulate cortex (ACC). Levels are measured in both resting and functional states using Magnetic Resonance Spectroscopy (MRS).
Change from Baseline in Inhibitory Control Performance | Baseline, Post-treatment (Week 12)
  Change from baseline to Week 12 in inhibitory control performance, as measured by the error rate on a Go-Nogo task. A decrease in the error rate indicates improvement.

SECONDARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale | Baseline, Week 4, Week 8, Week 12
  Change in the total score of the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) from baseline. Scores range from 0 to 40, with higher scores indicating greater symptom severity.
Yale-Brown Obsessive Compulsive Scale modified for Neurotic Excoriation | Baseline, Week 4, Week 8, Week 12
  Proportion of participants achieving a predefined percentage reduction in the total score from baseline to post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Huirong Zheng, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Mental Health Center, Guangdong Provincial People's Hospital, GuangDong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT06956157/ICF_001.pdf